CLINICAL TRIAL: NCT01667692
Title: Comparison of Azithromycin or Clarithromycin in 3drugs Protocol of H-pylori Eradication Regimen
Brief Title: Aizthromycin or Clarithromycin in H-pylori Eradication Regimen
Acronym: H-pylori
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shahid Sadoughi University of Medical Sciences and Health Services (Other)
Responsible Party: Principal Investigator, Behnam Baghianimoghadam, research consultant, Shahid Sadoughi University of Medical Sciences and Health Services
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ssu.hakimi-89027
Record Dates: First submitted 2012-08-12; First posted 2012-08-17 (Estimated); Last update posted 2012-08-17 (Estimated); Status verified 2012-08

CONDITIONS: Peptic Ulcer; Dyspepsia; H-pylori
Keywords: H-pylori; eradication; azithromycin; clarithromycin
MeSH Terms: conditions — Peptic Ulcer; Dyspepsia | interventions — Azithromycin; Clarithromycin

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- azithromycin (Experimental): Azithromycin (Zithromax, Azithrocin ) is an azalide, a subclass of macrolide antibiotics. Azithromycin is one of the world's best-selling antibiotics. It is derived from erythromycin, with a methyl-substituted nitrogen atom incorporated into the lactone ring, thus making the lactone ring 15-membered.
  Interventions: Drug: azithromycin
- clarithromycin (Experimental): Clarithromycin is a macrolide antibiotic used to treat pharyngitis, tonsillitis, acute maxillary sinusitis, acute bacterial exacerbation of chronic bronchitis, pneumonia (especially atypical pneumonias associated with Chlamydophila pneumoniae), skin and skin structure infections. In addition, it is sometimes used to treat legionellosis, Helicobacter pylori, and lyme disease.
  Interventions: Drug: clarithmycin

INTERVENTIONS:
Drug: azithromycin — Azithromycin (Zithromax, Azithrocin ) is an azalide, a subclass of macrolide antibiotics. Azithromycin is one of the world's best-selling antibiotics.[1] It is derived from erythromycin, with a methyl-substituted nitrogen atom incorporated into the lactone ring, thus making the lactone ring 15-membered.
  Other Names: (Zithromax, Azithrocin
  Arms: azithromycin
Drug: clarithmycin — Clarithromycin is a macrolide antibiotic used to treat pharyngitis, tonsillitis, acute maxillary sinusitis, acute bacterial exacerbation of chronic bronchitis, pneumonia (especially atypical pneumonias associated with Chlamydophila pneumoniae), skin and skin structure infections. In addition, it is sometimes used to treat legionellosis, Helicobacter pylori, and lyme disease.
  Other Names: Crixan, Claritt, Clarac, Biaxin, Klaricid, Klacid...
  Arms: clarithromycin

SUMMARY:
The Aim of this study is comparison between two regimens containing clarithromycinand azithromycin.

DETAILED DESCRIPTION:
Eradication of helicobacter pylori is important for treatment of GU but ideal regimen is not available.

HP is resistant to metronidazole and clarithromycin, thus clarithromycin is expensive and it is not available in underdevelopment countries.

There are different articles about replacement clarithromycin with azithromycin as a method of eradication of HP that is decreases length of therapy and increases, effectiveness of drugs and decreases resistance of drugs.

The Aim of this study is comparison between two regimens containing clarithromycinand azithromycin.

ELIGIBILITY:
Inclusion Criteria:

* patients with peptic ulcer due to H-pylori confirmed endoscopy and biopsy

Exclusion Criteria:

* patients who got H-pylori eradication treatment previously
* patients who used study drugs during 3months before study

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2011-03; Primary Completion 2011-11 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
H-pylori cinfirmation | 1-3 months before study
  confirmation is by endoscopy and biopsy

SECONDARY OUTCOMES:
h-pylori eradication confirmation | two months after completion of 14 days standard treatment
  confirmation of eradication was by endoscopy and biopsy
side effect of study srugs | during 14 days standard treatment
  it was assessed by researcher and self report of patients. variables like nausea, vomiting and diarrhea. the prevalence of each treatment related complain was registered by taking history from patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Behnam Baghianimoghadam, Yazd, Yazd Province, Iran